CLINICAL TRIAL: NCT05033288
Title: Prospective Comparative Effectiveness Trial of Carbon Ion Therapy, Surgery, and Proton Therapy for the Management of Pelvic Sarcomas (Soft Tissue/Bone) Involving the Bone
Brief Title: Comparing Carbon Ion Therapy, Surgery, and Proton Therapy for Management of Pelvic Sarcomas Involving the Bone
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC210709; NCI-2021-08847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC210709 (Other: Mayo Clinic); 21-004080 (Other: Mayo Clinic Institutional Review Board); ROF2181 (Other: Mayo Clinic Radiation Oncology)
Record Dates: First submitted 2021-08-23; First posted 2021-09-02 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Bone Sarcoma; Chondrosarcoma; Chordoma; Ewing Sarcoma of Bone; Pelvic Rhabdomyosarcoma
MeSH Terms: conditions — Bone Neoplasms; Chondrosarcoma; Chordoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational (questionnaires, medical record review): Patients complete quality of life questionnaires over 20 minutes at baseline (before any therapy), 2-4 and 5-9 months after completion of therapy, and then annually for up to 5 years. Patients' medical records are also reviewed.
  Interventions: Other: Electronic Health Record Review; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records are reviewed
Other: Quality-of-Life Assessment — Complete quality of life questionnaires
  Other Names: Quality of Life Assessment

SUMMARY:
This study compares carbon ion therapy, surgery, and proton therapy to determine if one has better disease control and fewer side effects. There are three types of radiation treatment used for pelvic bone sarcomas: surgery with or without photon/proton therapy, proton therapy alone, and carbon ion therapy alone. The purpose of this study is to compare quality of life among patients treated for pelvic bone sarcomas across the world, and to determine if carbon ion therapy improves quality of life compared to surgery and disease control compared with proton therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate whether carbon ion therapy provides improved patient reported health related quality of life (PRO-HRQOL) outcomes and less significant toxicities compared with surgery.

II. Demonstrate whether carbon ion therapy provides improved local control versus proton therapy.

OUTLINE:

Patients complete quality of life questionnaires over 20 minutes at baseline (before any therapy), 2-4 and 5-9 months after completion of therapy, and then annually for up to 5 years. Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Males and females >= 15 years of age
* Newly diagnosed, histologic confirmation of pelvic chordoma, chondrosarcoma, osteosarcoma, Ewing sarcoma with bone involvement, rhabdomyosarcoma (RMS) with bone involvement or non-RMS soft tissue sarcoma with bone involvement
* No evidence of distant sarcoma metastases as determined by clinical examination and any form of imaging
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Patients capable of childbearing must agree to use adequate contraception
* Ability to complete questionnaire(s) by themselves or with assistance
* Ability to provide written informed consent
* Chemotherapy per institutional guidelines is allowed

Exclusion Criteria:

* Patients receiving palliative treatment
* Recurrent disease
* Males and females < 15 years of age
* Previous radiation therapy to the site of the sarcoma or area surrounding it such that it would be partially or completely encompassed by the radiation volume needed to treat the current sarcoma. In other words, treatment on this study would require re-irradiation of tissues
* Patients with distant sarcoma metastases
* Benign pelvic bone histologies
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with newly diagnosed, histologic confirmation of pelvic chordoma, chondrosarcoma, osteosarcoma, Ewing sarcoma with bone involvement, rhabdomyosarcoma (RMS) with bone involvement or non-RMS soft tissue sarcoma with bone involvement treated with curative intent carbon ion radiation therapy (CIRT) at one of the carbon ion facilities in Europe or Asia or deemed appropriate to undergo definitive treatment with surgery or radiation therapy at Mayo Clinic (Minnesota, Florida, Arizona)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Average difference in change of functional quality of life (QOL) | Baseline (pre-treatment) to 1 year after completion of treatment
  Will be compared between patients who received carbon ion radiation therapy (CIRT) and surgery utilizing a one-sided test for a two sample t-test for independent means. The Patient Reported Outcomes Measurement Information System (PROMIS)-29 functional score will be calculated and median, mean, and 95% confidence interval will be computed for each arm, with one-sided two-sample t-tests conducted between the surgery +/- radiation therapy (RT) and CIRT arm.
Proportion of patients experiencing local control | Up to 5 years after completion of treatment
  Will be calculated along with 95% confidence intervals with a one-sided test for non-inferiority to be conducted between the PT and CIRT arms.
Progression-free survival - local control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including local control as well as progression-free survival for each arm and stratified by arm.
Progression-free survival - regional control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including regional control as well as progression-free survival for each arm and stratified by arm.
Progression-free survival - distant control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including distant control as well as progression-free survival for each arm and stratified by arm.
Overall survival - local control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including local control as well as overall survival for each arm and stratified by arm.
Overall survival - regional control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including regional control as well as overall survival for each arm and stratified by arm.
Overall survival - distant control | Up to 5 years after completion of treatment
  The Kaplan-Meier method with likelihood ratio tests will be used to calculate clinical outcomes including distant control as well as overall survival for each arm and stratified by arm.

SECONDARY OUTCOMES:
Secondary and exploratory analyses on toxicity data | Up to 5 years after completion of treatment
  Secondary and exploratory analyses on data will be conducted utilizing standard logistic regression analysis for acute (< 6 months) and late (> 6 months) toxicity.
Secondary and exploratory analyses on dose volume histogram (DVH) data | Up to 5 years after completion of treatment
  Secondary and exploratory analyses on data will be conducted utilizing standard logistic regression analysis for acute (< 6 months) and late (> 6 months) toxicity.
Dose volume histogram | Up to 5 years after completion of treatment
  Secondary and exploratory analyses on toxicity and DVH data will be conducted utilizing standard logistic regression analysis for acute (< 6 months) and late (> 6 months) toxicity. Receiver-operator curves and area-under-the curve will be computed separately for each DVH metric to determine the effect on toxicity, QOL, local control and survival.

CONTACTS AND LOCATIONS:
Overall Officials: Bradford S. Hoppe, MD, MPH, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials